CLINICAL TRIAL: NCT03272100
Title: Influence of Two Different Flap Designs for Sinus Floor Elevation. A Split-mouth Randomised Controlled Clinical Trial
Brief Title: Influence of Two Different Flap Designs for Sinus Floor Elevation
Status: Completed | Type: Observational
Sponsor: University of Firenze and Siena, Napoli, Italy (Other)
Responsible Party: Principal Investigator, nicola baldini, principal investigator, University of Firenze and Siena, Napoli, Italy
Other Study IDs: MSL001
Record Dates: First submitted 2017-08-24; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Bone Involvement in Diseases Classified Elsewhere
Keywords: lateral approach; bone augmentation; sinus lift; flap
MeSH Terms: interventions — Surgical Flaps; Sinus Floor Augmentation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test side ( horizontal flap): Horizontal incision was realised in alveolar mucosa, in order to obtain the exposure of the lateral wall of the maxillary sinus, thus accessing the sinus cavity
  Interventions: Procedure: flap
- control side ( standard flap): Trapezoidal flap was realised, using a crestal incision and two deep vertical incisions extended in the fornix to expose the lateral wall of the maxillary sinus
  Interventions: Procedure: flap

INTERVENTIONS:
Procedure: flap — after flap incision , the sinus cavity was opened and then the membrane raised up
  Other Names: surgical approach; Sinus augmentation

SUMMARY:
It is assumed that the reduction of the flap dimension could provide a reduction of surgical time, post surgical complications and patient's discomfort when compared with the traditional surgical approach.

DETAILED DESCRIPTION:
16 edentulous patients in maxillary posterior area were treated with a bilateral sinus lift procedure. Once enrolled in the study impressions were realised and the radiographic stent prepared, with radio-opaque references fixed in the positions where the implants should be inserted. Pre-surgical CT scan was executed after placing the stent in its proper position in patient's mouth. If no surgical contra-indications were detected at CT evaluation, patients were involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* patient edentulous in the maxillary posterior area on both left and right side
* residual bone height in the maxillary premolar and molar region less than 4mm

Exclusion Criteria:

* history of systemic diseases that would contraindicate surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all the involved patients were edentulous in the maxillary posterior area , bilaterally, with a residual bone heigh of less then 4 mm; for this reason they required a surgical bone reconstruction for implant placement.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
height of augmented bone obtained | 6 months
  the height of the gained bone was recorded by using the control CT scan, realized after 6 months of follow up

SECONDARY OUTCOMES:
Duration of the surgery | 1 day
  both total and partial times of different surgical steps were recorded
Post surgical patient's discomfort | 2 weeks
  all patients were asked to fill out a VAS scale, graduated from 1 (minimal pain ) to 10 ( maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: marco ferrari, clinical director, Study Chair — tuscan school of dental medicine, university of Firenze and Siena
Locations (2):
- Italy (2):
  - Siena University, Department of Periodontology, Policlinico Le Scotte Siena., Siena
  - Tuscan School of Dentistry, Siena